CLINICAL TRIAL: NCT00968539
Title: Safety and Immunogenicity Study of GSK Biologicals' Influenza Vaccine GSK2340272A in Adults Aged 18 to 60 Years
Brief Title: Study to Evaluate the Immunogenicity & Safety of an Investigational Influenza Vaccine (H1N1) in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 113456; 2009-013710-27 (EudraCT Number)
Record Dates: First submitted 2009-08-27; First posted 2009-08-31 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Influenza
Keywords: GSK Bio's influenza vaccine GSK2340272A; influenza infection
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- GSK2340272A GROUP (Experimental): Healthy male or female adults, between and including 18 to 60 years of age, who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
  Interventions: Biological: GSK investigational vaccine GSK2340272A
- GSK2340269A GROUP (Experimental): Healthy male or female adults, between and including 18 to 60 years of age, who received two doses of GSK2340269A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
  Interventions: Biological: GSK investigational vaccine GSK2340269A

INTERVENTIONS:
Biological: GSK investigational vaccine GSK2340272A — Two intramuscular injections
  Arms: GSK2340272A GROUP
Biological: GSK investigational vaccine GSK2340269A — Two intramuscular injections
  Arms: GSK2340269A GROUP

SUMMARY:
The objective of the study is to evaluate the immunogenicity and safety of GSK Biologicals' investigational vaccine GSK2340272A.

ELIGIBILITY:
Inclusion Criteria:

* A male or female aged 18 to 60 years at the time of the first vaccination.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol
* Written informed consent obtained from the subject.
* Satisfactory baseline medical assessment by history and physical examination. Stable health status is defined as the absence of health event satisfying the definition of a serious adverse event, or a change in an ongoing drug therapy due to therapeutic failure or symptoms of drug toxicity, within one month prior to enrollment.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or multiple-user device.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:
* has practiced adequate contraception for 30 days prior to vaccination, and
* has a negative pregnancy test on the day of vaccination, and
* has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period. Potential subjects in the follow-up phase of a prior investigational study may be enrolled if the investigator's judgment is that it will have no effect on safety, reactogenicity, or immunogenicity endpoints in this study, and that it does not violate the protocol requirements of the prior trial.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of an axillary temperature >= 37.5°C, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination. NOTE: The subject may be vaccinated at a later date, provided symptoms have resolved, vaccination occurs within the window specified by the protocol, and all other eligibility criteria continue to be satisfied.
* Diagnosed with cancer, or treatment for cancer, within the past 3 years.
* Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.
* Persons with a history of histological-confirmed basal cell carcinoma of the skin successfully treated with local excisions only are excepted and may enroll within 3 years of diagnosis, but other histological types of skin cancer require a 3-year untreated and disease-free window as above.
* Women who are disease free 3 years or more after the treatment for breast cancer and receiving long-term prophylactic tamoxifen are excepted and may enroll.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Clinically or virologically confirmed influenza infection within 6 months preceding the study start.
* Chronic administration of immunosuppressants or other immune modifying drugs within 6 months of study enrolment or planned administration during the study period.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrolment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose aspirin, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome.
* Administration of any vaccines within 30 days before vaccination.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* Pregnant or lactating female
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any conditions which, in the opinion of the investigator, prevents the subjects from participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2009-09-08 (Actual); Primary Completion 2010-09-28 (Actual); Study Completion 2010-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Roman F, Clement F, Dewe W, Walravens K, Maes C, Willekens J, De Boever F, Hanon E, Leroux-Roels G. Effect on cellular and humoral immune responses of the AS03 adjuvant system in an A/H1N1/2009 influenza virus vaccine administered to adults during two randomized controlled trials. Clin Vaccine Immunol. 2011 May;18(5):835-43. doi: 10.1128/CVI.00480-10. Epub 2011 Mar 30. PMID 21450978
- [Derived] van der Most RG, Clement F, Willekens J, Dewe W, Walravens K, Vaughn DW, Leroux-Roels G. Long-Term Persistence of Cell-Mediated and Humoral Responses to A(H1N1)pdm09 Influenza Virus Vaccines and the Role of the AS03 Adjuvant System in Adults during Two Randomized Controlled Trials. Clin Vaccine Immunol. 2017 Jun 5;24(6):e00553-16. doi: 10.1128/CVI.00553-16. Print 2017 Jun. PMID 28446441
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 113456 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113456 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113456 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113456 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113456 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113456 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113456 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK2340272A Group | GSK2340269A Group
Started | 64 | 66
Completed | 63 | 66
Not Completed | 1 | 0
Not completed — Lost to follow-up (incompl. vaccination) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2340272A Group | GSK2340269A Group | Total
Number analyzed (Participants) | 64 | 66 | 130
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.1 (13.53) | 38.2 (14.10) | 38.64 (13.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 39 | 80
  Male | 23 | 27 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-East Asian heritage | 0 | 1 | 1
  White-Caucasian/European heritage | 64 | 65 | 129

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Hemagglutination Inhibition (HI) Antibodies
Description: Seroconversion was defined as: For initially seronegative subjects [antibody titer below (<) 1:10 prior to vaccination], antibody titer greater than or equal to (≥) 1:40 after vaccination; For initially seropositive subjects (antibody titer ≥ 1:10 prior to vaccination), antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was A/California/7/2009 (H1N1)v-like influenza (Flu A/CAL/7/09).
Time Frame: At Day 42
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects who received 2 vaccine doses and for whom assay results were available for antibodies against H1N1 antigen for the blood sample taken up to 21 days after the second vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group
Number analyzed (Participants) | 59
Participants | 58

2. Primary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: A seroprotected subject was defined as a vaccinated subject with a serum hemagglutination inhibition (HI) titer ≥ 1:40. The flu strain assessed was A/California/7/2009 (H1N1)v-like influenza (Flu A/CAL/7/09).
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group
Number analyzed (Participants) | 59
Participants | 59

3. Primary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: GMFR, also called seroconversion factor (SCF), was defined as the fold increase in serum HI geometric mean titers (GMTs) post-vaccination compared to pre-vaccination. The flu strain assessed was Flu A/CAL/7/09.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340272A Group
Number analyzed (Participants) | 59
Fold increase | 72.9 [55.4 to 95.9]

4. Secondary Outcome: Number of Subjects With HI Antibody Concentrations Above the Cut-off Value
Description: Seropositivity cut-off values assessed were equal to or above (≥) 1:10 in the sera of subjects seronegative before vaccination. The Flu strain assessed was Flu A/CAL/7/09.
Time Frame: At Days 0, 21 and 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 60 | 66
Participants
  Flu A/CAL/7/09, Day 0 | 23 | 28
  Flu A/CAL/7/09, Day 21 | 60 | 65
  Flu A/CAL/7/09, Day 42: number analyzed (Participants) | 59 | 66
  Flu A/CAL/7/09, Day 42 | 59 | 66

5. Secondary Outcome: Number of Subjects With HI Antibody Concentrations Above the Cut-off Value
Description: as for outcome 4
Time Frame: At Day 182
Population: The analysis was performed on the ATP cohort for persistence at Month 6, which included all evaluable subjects for whom assay results were available for antibodies against the study vaccine antigen component at Month 6.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 59 | 61
Participants | 59 | 61

6. Secondary Outcome: Number of Subjects With HI Antibody Concentrations Above the Cut-off Value
Description: Seropositivity cut-off values assessed were equal to or above (≥) 1:10 in the sera of subjects seronegative before vaccination. The Flu strain assessed was Flu A/CAL/09.
Time Frame: At Day 364
Population: The analysis was performed on the ATP cohort for persistence at Month 12, which included all evaluable subjects who met all eligibility criteria and for whom assay results were available for antibodies against the study vaccine antigen component at Month 12.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 59 | 65
Participants | 59 | 62

7. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The flu strain assessed was Flu A/CAL/7/09. The reference seropositivity cut-off value was ≥ 1:10.
Time Frame: At Days 0, 21 and 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 60 | 66
Titers
  Flu A/CAL/7/09, Day 0 | 8.8 [7.0 to 11.1] | 10.8 [8.1 to 14.4]
  Flu A/CAL/7/09, Day 21 | 335.2 [250.1 to 449.2] | 310.2 [218.8 to 439.7]
  Flu A/CAL/7/09, Day 42: number analyzed (Participants) | 59 | 66
  Flu A/CAL/7/09, Day 42 | 636.3 [520.9 to 777.3] | 341.0 [259.9 to 447.3]

8. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 7
Time Frame: At Day 182
Population: The analysis was performed on the ATP cohort for persistence at Month 6, which included all evaluable subjects who met all eligibility criteria and for whom assay results were available for antibodies against the study vaccine antigen component at Month 6.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 59 | 61
Titers | 204.8 [161.5 to 259.8] | 146.1 [108.5 to 196.7]

9. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 7
Time Frame: At Day 364
Population: The analysis was performed on the ATP cohort for persistence at Month 12, which included all evaluable subjects for whom assay results were available for antibodies against the study vaccine antigen component at Month 12.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 59 | 65
Titers | 85.8 [64.4 to 114.3] | 87.6 [64.7 to 118.8]

10. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies
Description: Seroconversion was defined as: For initially seronegative subjects (antibody titer < 1:10 prior to vaccination), antibody titer ≥ 1:40 after vaccination; For initially seropositive subjects (antibody titer ≥ 1:10 prior to vaccination), antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was A/California/7/2009 (H1N1)v-like influenza (Flu A/CAL/7/09).
Time Frame: At Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 60 | 66
Participants | 59 | 56

11. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies
Description: as for outcome 10
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340269A Group
Number analyzed (Participants) | 66
Participants | 61

12. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies
Description: as for outcome 10
Time Frame: At Day 182
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 59 | 61
Participants | 57 | 47

13. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies
Description: as for outcome 10
Time Frame: At Day 364
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 59 | 65
Participants | 41 | 46

14. Secondary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: as for outcome 2
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 60 | 66
Participants
  Flu A/CAL/7/09, Day 0 | 7 | 12
  Flu A/CAL/7/09, Day 21 | 60 | 62

15. Secondary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: as for outcome 2
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340269A Group
Number analyzed (Participants) | 66
Participants | 66

16. Secondary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: as for outcome 2
Time Frame: At Day 182
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 59 | 61
Participants | 59 | 52

17. Secondary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: as for outcome 2
Time Frame: At Day 364
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 59 | 65
Participants | 46 | 55

18. Secondary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: Seroconversion factor (SCF) was defined as the fold increase in serum HI geometric mean titers (GMTs) post-vaccination compared to pre-vaccination. The flu strain assessed was Flu A/CAL/7/09.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 60 | 66
Fold increase | 38.1 [28.6 to 50.7] | 28.7 [20.0 to 41.2]

19. Secondary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 18
Time Frame: At Day 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340269A Group
Number analyzed (Participants) | 66
Fold increase | 31.5 [23.1 to 43.2]

20. Secondary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 18
Time Frame: At Day 182
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 59 | 61
Fold increase | 22.5 [18.0 to 28.2] | 13.9 [10.2 to 18.9]

21. Secondary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 18
Time Frame: At Day 364
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 59 | 65
Fold increase | 9.7 [7.4 to 12.5] | 8.3 [6.2 to 11.0]

22. Secondary Outcome: Titers for Serum Neutralizing Antibodies Against Flu A/Neth/602/09 Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The flu strain assessed was Flu A/Neth/602/09. The reference seropositivity cut-off value was ≥ 1:8.
Time Frame: At Days 0, 21 and 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 28 | 30
Titers
  Flu A/Neth/602/09, Day 0 | 6.1 [4.6 to 8.0] | 9.6 [6.7 to 13.6]
  Flu A/Neth/602/09, Day 21 | 152.3 [78.4 to 295.9] | 89.9 [51.6 to 156.6]
  Flu A/Neth/602/09, Day 42 | 243.8 [163.4 to 363.7] | 144.9 [88.7 to 236.6]

23. Secondary Outcome: Number of Seroconverted Subjects for Serum Neutralizing Antibodies Against Flu A/Neth/602/09
Description: Seroconversion was defined as: For initially seronegative subjects, antibody titer ≥ 1:32 after vaccination; For initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was Flu A/Neth/602/09.
Time Frame: At Days 21 and 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 28 | 30
Participants
  Flu A/Neth/602/09, Day 21 | 21 | 22
  Flu A/Neth/602/09, Day 42 | 27 | 23

24. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with the symptom sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 63 | 66
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 63 | 65
  Any Pain, Dose 1 | 57 | 23
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 63 | 65
  Grade 3 Pain, Dose 1 | 1 | 0
  Any Redness, Dose 1: number analyzed (Participants) | 63 | 65
  Any Redness, Dose 1 | 1 | 0
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 63 | 65
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1: number analyzed (Participants) | 63 | 65
  Any Swelling, Dose 1 | 5 | 0
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 63 | 65
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 62 | 66
  Any Pain, Dose 2 | 56 | 20
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 62 | 66
  Grade 3 Pain, Dose 2 | 2 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 62 | 66
  Any Redness, Dose 2 | 3 | 0
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 62 | 66
  Grade 3 Redness, Dose 2 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 62 | 66
  Any Swelling, Dose 2 | 9 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 62 | 66
  Grade 3 Swelling, Dose 2 | 0 | 0
  Any Pain, Across Doses | 61 | 32
  Grade 3 Pain, Across Doses | 3 | 0
  Any Redness, Across Doses | 4 | 0
  Grade 3 Redness, Across Doses | 0 | 0
  Any Swelling, Across Doses | 11 | 0
  Grade 3 Swelling, Across Doses | 0 | 0

25. Secondary Outcome: Number of Days With Solicited Local Symptoms
Description: The number of days with any solicited local symptoms reported during the solicited post-vaccination period. There were no subjects from GSK2340269A Group who reported Redness or Swelling.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects with the symptom sheet filled in.
Measure: Median (Inter-Quartile Range); unit: Days
Units Other Than Participants: Doses with the symptom
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 63 | 66
Number analyzed (Doses with the symptom) | 113 | 43
Days
  Pain, post-Dose 1: number analyzed (Participants) | 63 | 65
  Pain, post-Dose 1: number analyzed (Doses with the symptom) | 57 | 23
  Pain, post-Dose 1 | 3.0 [2.0 to 4.0] | 1.0 [1.0 to 2.0]
  Pain, post-Dose 2: number analyzed (Participants) | 62 | 66
  Pain, post-Dose 2: number analyzed (Doses with the symptom) | 56 | 20
  Pain, post-Dose 2 | 3.0 [2.0 to 4.0] | 2.0 [1.0 to 3.0]
  Pain, Overall/dose | 3.0 [2.0 to 4.0] | 2.0 [1.0 to 2.0]
  Redness, post-Dose 1: number analyzed (Participants) | 63 | 65
  Redness, post-Dose 1: number analyzed (Doses with the symptom) | 1 | 0
  Redness, post-Dose 1 | 3.0 [3.0 to 3.0] |
  Redness, post-Dose 2: number analyzed (Participants) | 62 | 66
  Redness, post-Dose 2: number analyzed (Doses with the symptom) | 3 | 0
  Redness, post-Dose 2 | 2.0 [2.0 to 3.0] |
  Redness, Overall/dose: number analyzed (Doses with the symptom) | 4 | 0
  Redness, Overall/dose | 2.5 [2.0 to 3.0] |
  Swelling, post-Dose 1: number analyzed (Participants) | 63 | 65
  Swelling, post-Dose 1: number analyzed (Doses with the symptom) | 5 | 0
  Swelling, post-Dose 1 | 2.0 [2.0 to 2.0] |
  Swelling, post-Dose 2: number analyzed (Participants) | 62 | 66
  Swelling, post-Dose 2: number analyzed (Doses with the symptom) | 9 | 0
  Swelling, post-Dose 2 | 2.0 [2.0 to 2.0] |
  Swelling, Overall/dose: number analyzed (Doses with the symptom) | 14 | 0
  Swelling, Overall/dose | 2.0 [2.0 to 2.0] |

26. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were Fatigue, Headache, Joint pain at other location, Muscle aches, Shivering, Sweating and Fever [defined as axillary temperature equal to or above ≥ 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = temperature > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 63 | 66
Participants
  Any Fatigue, Dose 1: number analyzed (Participants) | 63 | 65
  Any Fatigue, Dose 1 | 22 | 18
  Grade 3 Fatigue, Dose 1: number analyzed (Participants) | 63 | 65
  Grade 3 Fatigue, Dose 1 | 0 | 1
  Related Fatigue, Dose 1: number analyzed (Participants) | 63 | 65
  Related Fatigue, Dose 1 | 21 | 16
  Any Headache, Dose 1: number analyzed (Participants) | 63 | 65
  Any Headache, Dose 1 | 17 | 11
  Grade 3 Headache, Dose 1: number analyzed (Participants) | 63 | 65
  Grade 3 Headache, Dose 1 | 1 | 0
  Related Headache, Dose 1: number analyzed (Participants) | 63 | 65
  Related Headache, Dose 1 | 15 | 8
  Any Joint pain, Dose 1: number analyzed (Participants) | 63 | 65
  Any Joint pain, Dose 1 | 7 | 4
  Grade 3 Joint pain, Dose 1: number analyzed (Participants) | 63 | 65
  Grade 3 Joint pain, Dose 1 | 0 | 0
  Related Joint pain, Dose 1: number analyzed (Participants) | 63 | 65
  Related Joint pain, Dose 1 | 7 | 3
  Any Muscle aches, Dose 1: number analyzed (Participants) | 63 | 65
  Any Muscle aches, Dose 1 | 20 | 6
  Grade 3 Muscle aches, Dose 1: number analyzed (Participants) | 63 | 65
  Grade 3 Muscle aches, Dose 1 | 1 | 0
  Related Muscle aches, Dose 1: number analyzed (Participants) | 63 | 65
  Related Muscle aches, Dose 1 | 20 | 4
  Any Shivering, Dose 1: number analyzed (Participants) | 63 | 65
  Any Shivering, Dose 1 | 6 | 4
  Grade 3 Shivering, Dose 1: number analyzed (Participants) | 63 | 65
  Grade 3 Shivering, Dose 1 | 0 | 1
  Related Shivering, Dose 1: number analyzed (Participants) | 63 | 65
  Related Shivering, Dose 1 | 6 | 2
  Any Sweating, Dose 1: number analyzed (Participants) | 63 | 65
  Any Sweating, Dose 1 | 6 | 7
  Grade 3 Sweating, Dose 1: number analyzed (Participants) | 63 | 65
  Grade 3 Sweating, Dose 1 | 0 | 0
  Related Sweating, Dose 1: number analyzed (Participants) | 63 | 65
  Related Sweating, Dose 1 | 6 | 5
  Any Fever, Dose 1: number analyzed (Participants) | 63 | 65
  Any Fever, Dose 1 | 0 | 0
  Grade 3 Fever, Dose 1: number analyzed (Participants) | 63 | 65
  Grade 3 Fever, Dose 1 | 0 | 0
  Related Fever, Dose 1: number analyzed (Participants) | 63 | 65
  Related Fever, Dose 1 | 0 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 62 | 66
  Any Fatigue, Dose 2 | 28 | 13
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 62 | 66
  Grade 3 Fatigue, Dose 2 | 2 | 2
  Related Fatigue, Dose 2: number analyzed (Participants) | 62 | 66
  Related Fatigue, Dose 2 | 27 | 13
  Any Headache, Dose 2: number analyzed (Participants) | 62 | 66
  Any Headache, Dose 2 | 22 | 9
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 62 | 66
  Grade 3 Headache, Dose 2 | 2 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 62 | 66
  Related Headache, Dose 2 | 20 | 8
  Any Joint pain, Dose 2: number analyzed (Participants) | 62 | 66
  Any Joint pain, Dose 2 | 13 | 4
  Grade 3 Joint pain, Dose 2: number analyzed (Participants) | 62 | 66
  Grade 3 Joint pain, Dose 2 | 0 | 0
  Related Joint pain, Dose 2: number analyzed (Participants) | 62 | 66
  Related Joint pain, Dose 2 | 13 | 4
  Any Muscle aches, Dose 2: number analyzed (Participants) | 62 | 66
  Any Muscle aches, Dose 2 | 23 | 7
  Grade 3 Muscle aches, Dose 2: number analyzed (Participants) | 62 | 66
  Grade 3 Muscle aches, Dose 2 | 2 | 0
  Related Muscle aches, Dose 2: number analyzed (Participants) | 62 | 66
  Related Muscle aches, Dose 2 | 23 | 6
  Any Shivering, Dose 2: number analyzed (Participants) | 62 | 66
  Any Shivering, Dose 2 | 11 | 3
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 62 | 66
  Grade 3 Shivering, Dose 2 | 0 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 62 | 66
  Related Shivering, Dose 2 | 11 | 2
  Any Sweating, Dose 2: number analyzed (Participants) | 62 | 66
  Any Sweating, Dose 2 | 12 | 7
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 62 | 66
  Grade 3 Sweating, Dose 2 | 1 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 62 | 66
  Related Sweating, Dose 2 | 12 | 6
  Any Fever, Dose 2: number analyzed (Participants) | 62 | 66
  Any Fever, Dose 2 | 2 | 0
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 62 | 66
  Grade 3 Fever, Dose 2 | 0 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 62 | 66
  Related Fever, Dose 2 | 2 | 0
  Any Fatigue, Across doses | 34 | 22
  Grade 3 Fatigue, Across doses | 2 | 3
  Related Fatigue, Across doses | 33 | 22
  Any Headache, Across doses | 29 | 14
  Grade 3 Headache, Across doses | 3 | 0
  Related Headache, Across doses | 27 | 12
  Any Joint pain, Across doses | 14 | 6
  Grade 3 Joint pain, Across doses | 0 | 0
  Related Joint pain, Across doses | 14 | 6
  Any Muscle aches, Across doses | 27 | 12
  Grade 3 Muscle aches, Across doses | 3 | 0
  Related Muscle aches, Across doses | 27 | 10
  Any Shivering, Across doses | 14 | 6
  Grade 3 Shivering, Across doses | 0 | 1
  Related Shivering, Across doses | 14 | 4
  Any Sweating, Across doses | 14 | 11
  Grade 3 Sweating, Across doses | 1 | 0
  Related Sweating, Across doses | 14 | 9
  Any Fever, Across doses | 2 | 0
  Grade 3 Fever, Across doses | 0 | 0
  Related Fever, Across doses | 2 | 0

27. Secondary Outcome: Number of Days With Solicited General Symptoms
Description: The number of days with any solicited general symptoms reported during the solicited post-vaccination period. There were no subjects from GSK2340269A Group who reported Temperature.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 24
Measure: Median (Inter-Quartile Range); unit: Days
Units Other Than Participants: Doses with the symptom
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 63 | 66
Number analyzed (Doses with the symptom) | 50 | 31
Days
  Fatigue, post-Dose 1: number analyzed (Participants) | 63 | 65
  Fatigue, post-Dose 1: number analyzed (Doses with the symptom) | 22 | 18
  Fatigue, post-Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0]
  Fatigue, post-Dose 2: number analyzed (Participants) | 62 | 66
  Fatigue, post-Dose 2: number analyzed (Doses with the symptom) | 28 | 13
  Fatigue, post-Dose 2 | 1.5 [1.0 to 3.0] | 3.0 [2.0 to 4.0]
  Fatigue, Overall/dose | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Headache, post-Dose 1: number analyzed (Participants) | 63 | 65
  Headache, post-Dose 1: number analyzed (Doses with the symptom) | 17 | 11
  Headache, post-Dose 1 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]
  Headache, post-Dose 2: number analyzed (Participants) | 62 | 66
  Headache, post-Dose 2: number analyzed (Doses with the symptom) | 22 | 9
  Headache, post-Dose 2 | 2.0 [1.0 to 2.0] | 2.0 [2.0 to 3.0]
  Headache, Overall/dose: number analyzed (Doses with the symptom) | 39 | 20
  Headache, Overall/dose | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Joint pain, post-Dose 1: number analyzed (Participants) | 63 | 65
  Joint pain, post-Dose 1: number analyzed (Doses with the symptom) | 7 | 4
  Joint pain, post-Dose 1 | 3.0 [1.0 to 4.0] | 2.0 [1.5 to 3.0]
  Joint pain, post-Dose 2: number analyzed (Participants) | 62 | 66
  Joint pain, post-Dose 2: number analyzed (Doses with the symptom) | 13 | 4
  Joint pain, post-Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.5]
  Joint pain, Overall/dose: number analyzed (Doses with the symptom) | 20 | 8
  Joint pain, Overall/dose | 1.5 [1.0 to 3.0] | 2.0 [1.0 to 3.5]
  Muscle aches, post-Dose 1: number analyzed (Participants) | 63 | 65
  Muscle aches, post-Dose 1: number analyzed (Doses with the symptom) | 20 | 6
  Muscle aches, post-Dose 1 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Muscle aches, post-Dose 2: number analyzed (Participants) | 62 | 66
  Muscle aches, post-Dose 2: number analyzed (Doses with the symptom) | 23 | 7
  Muscle aches, post-Dose 2 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]
  Muscle aches, Overall/dose: number analyzed (Doses with the symptom) | 43 | 13
  Muscle aches, Overall/dose | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Sweating, post-Dose 1: number analyzed (Participants) | 63 | 65
  Sweating, post-Dose 1: number analyzed (Doses with the symptom) | 6 | 7
  Sweating, post-Dose 1 | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0]
  Sweating, post-Dose 2: number analyzed (Participants) | 62 | 66
  Sweating, post-Dose 2: number analyzed (Doses with the symptom) | 12 | 7
  Sweating, post-Dose 2 | 1.5 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Sweating, Overall/dose: number analyzed (Doses with the symptom) | 18 | 14
  Sweating, Overall/dose | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Shivering, post-Dose 1: number analyzed (Participants) | 63 | 65
  Shivering, post-Dose 1: number analyzed (Doses with the symptom) | 6 | 4
  Shivering, post-Dose 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0]
  Shivering, post-Dose 2: number analyzed (Participants) | 62 | 66
  Shivering, post-Dose 2: number analyzed (Doses with the symptom) | 11 | 3
  Shivering, post-Dose 2 | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Shivering, Overall/dose: number analyzed (Doses with the symptom) | 17 | 7
  Shivering, Overall/dose | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0]
  Temperature, post-Dose 2: number analyzed (Participants) | 62 | 66
  Temperature, post-Dose 2: number analyzed (Doses with the symptom) | 2 | 0
  Temperature, post-Dose 2 | 2.0 [2.0 to 2.0] |
  Temperature, Overall/dose: number analyzed (Doses with the symptom) | 2 | 0
  Temperature, Overall/dose | 2.0 [2.0 to 2.0] |

28. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within 21 days after the first vaccination and 63 days after the second vaccination (Day 0 - Day 20 and Day 21 - Day 83)
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 64 | 66
Participants
  Any AE(s) | 39 | 38
  Grade 3 AE(s) | 7 | 9
  Related AE(s) | 12 | 7

29. Secondary Outcome: Number of Subjects With Adverse Events of Specific Interest (AESIs)
Description: An AESI was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration.
Time Frame: During the entire study period (from Day 0 up to Day 364)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 64 | 66
Participants | 1 | 1

30. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 0 up to Day 364)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 64 | 66
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: within the 84-day (Days 0-83) post-vaccination period; SAEs: during the entire study period (from Day 0 up to Day 364).
Description: The solicited local and general symptoms were only collected from those subjects who filled in their symptom sheets.
Arm/Group | GSK2340272A Group | GSK2340269A Group
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/66
Serious Adverse Events (participants affected / at risk) | 2/64 | 1/66
Other Adverse Events (participants affected / at risk) | 62/64 | 48/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2340272A Group (N=64) | GSK2340269A Group (N=66)
Migraine (Nervous system disorders) | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK2340272A Group (N=64) | GSK2340269A Group (N=66)
Pain (General disorders) | 61/63 | 32
Redness (General disorders) | 4/63 | 0
Swelling (General disorders) | 11/63 | 0
Fatigue (General disorders) | 34/63 | 22
Headache (General disorders) | 29/63 | 14
Joint pain (General disorders) | 14/63 | 6
Muscle aches (General disorders) | 27/63 | 12
Shivering (General disorders) | 14/63 | 6
Sweating (General disorders) | 14/63 | 11
Upper respiratory tract infection (Infections and infestations) | 6 | 11
Headache (Nervous system disorders) | 7 | 7
Rhinitis (Infections and infestations) | 10 | 3
Influenza like illness (General disorders) | 4 | 6
Nausea (Gastrointestinal disorders) | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.